CLINICAL TRIAL: NCT03302325
Title: Circulating Tumor DNA As Liquid Biopsy in Patients with Stage IV Solid Tumors, a Feasibility Study At MUSC HCC
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 102718
Record Dates: First submitted 2017-08-09; First posted 2017-10-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor, Adult
Keywords: stage IV solid tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — circulating tumor DNA (ctDNA) in the blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Stage IV solid tumors: adult patients with stage IV cancer that are starting a new line of treatment
  Interventions: Procedure: research blood draws

INTERVENTIONS:
Procedure: research blood draws — Twenty-five mL of peripheral blood (PB) will be collected for research. Blood will be collected in EDTA tubes and used to isolate ctDNA. For each subject we will request that he/she contribute 25 mL of plasma no more frequently than every 6 weeks, and at same time of standard of care blood draws and routine clinic visit, and for no more than 3 times (including baseline and end of study).

SUMMARY:
1. To demonstrate the ability to detect specific cancer mutations in ctDNA isolated from plasma of stage IV cancer patients at HCC.
2. To compare, in each patient, ctDNA longitudinal samples through treatment, and when available, with those of primary tumor and metastasis.

DETAILED DESCRIPTION:
The overall goal of this study is to study circulating tumor DNA (ctDNA) in the blood to determine how cancer cells in patients react to treatment. DNA is short for deoxyribonucleic acid. DNA contains information that determines in part the traits, such as eye color, height, or disease risk, that are passed on from parent to child. This reaction will be measured by studying patient blood that will be collected before and during treatment until there is disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of stage IV malignancy, including any advanced solid tumors (including lymphoma)
* Eastern Cooperative Oncology Group (ECOG) performance Status (PS) 0-3
* Life expectancy ≥ 3 months
* Patients must be able to provide consent
* Patients can be enrolled in other interventional clinical trials

Exclusion Criteria:

- Age < 18-year-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with stage IV cancer that start a new line of treatment and agree to have blood drawn
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Detecting specific cancer mutations in ctDNA isolated from plasma of stage IV cancer patients at HCC. | 24 months
Changes in patients' ctDNA longitudinal samples through treatment, and when available, of primary tumor and metastasis. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Giordano, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States